CLINICAL TRIAL: NCT03123822
Title: To Compare the Effectiveness of 3 Different Types of Lens and Lens Coating in Eliminating Symptoms for Children With Prolonged Visual Symptoms Due to a Concussion.
Brief Title: Spectacles Lens in Concussed Kids
Acronym: SLICK
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not enough interest/participants. Recruitment was more difficult due to pandemic
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Katherine K Weise, Director of Pediatric Optometry Services, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020
Record Dates: First submitted 2017-04-13; First posted 2017-04-21 (Actual); Results first posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-05

CONDITIONS: Concussion, Mild; Convergence Insufficiency; Accommodation; Insufficiency
MeSH Terms: conditions — Brain Concussion; Ocular Motility Disorders | interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Single vision glasses (Experimental): Typical glasses prescribed for children to correct only distance refractive error and to be worn all waking hours.
  Interventions: Device: Glasses
- Single vision glasses with anti-glare coating (Experimental): Typical glasses prescribed for children to correct only distance prescription with anti-glare coating and to be worn all waking hours.
  Interventions: Device: Glasses
- Eyezen (Experimental): Commercially available, low-powered, progressive addition lenses glasses with anti-glare coating to be worn all waking hours
  Interventions: Device: Glasses

INTERVENTIONS:
Device: Glasses — Glasses traditionally prescribed for refractive error

SUMMARY:
We will be looking at 3 treatment arms in the form of different type of glasses to see if one is superior to helping kids have sustained a concussion and are symptomatic.

DETAILED DESCRIPTION:
Recent studies have shown children who sustain a concussion are susceptible to having chronic symptoms (post-concussion syndrome). This chronicity can lead to delays in returning to learn and returning to play. Blurry vision, double vision, eye strain and eye tracking problems are some of the reported chronic symptoms that can affect patients' daily activities. Concussion awareness has increased recently and there is a surge of interest to better understand and treat the symptoms of post-concussion syndrome. Currently, ocular treatment for patients are often empirically determined. Common treatments are vision therapy and/or bifocal glasses. There has yet to be any standardization or prospective studies looking into treatment for these concussed patients with ocular symptoms and findings. The objective of this protocol is to compare three different types of glasses (typical prescription glasses for kids, typical glasses for kids with anti-glare coating, and progressive addition lenses with anti-glare coating) as treatment options for participants who are still symptomatic four weeks out from their concussion. The main outcome is the effectiveness of these three different options in reducing patients' symptoms and improving the participants' visual findings.

ELIGIBILITY:
Inclusion Criteria:

* Sustained a concussion > 6 weeks < 16 weeks from date of initial visit
* Criteria for concussion: formally diagnosed by physician
* Minimum best corrected visual acuity: 20/25 in right and left eyes at distance and 20/30 both eyes at near
* Minimum Stereopsis: 500" global
* CISS score > 16
* Refractive error at least + 0.50D sphere or cylinder
* Ability to clear > 0.50 cycles per minute in monocular accommodative flipper of and binocular accommodative flipper of +/-1.50

Exclusion Criteria:

* Diplopia from nerve palsies
* Retinal pathology
* Previous treatment of any amount of bifocal lenses and base in prism since concussion.
* Vision therapy > 6 weeks since concussion

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Becky Luu, OD, Study Director — University of Alabama at Birmingham; Katherine Weise, OD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama School of Optometry, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Vision Glasses | Single Vision Glasses With Anti-glare Coating | Eyezen
Started | 1 | 1 | 3
Completed | 1 | 1 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: It is not different from the assignment in participant flow
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Vision Glasses | Single Vision Glasses With Anti-glare Coating | Eyezen | Total
Number analyzed (Participants) | 1 | 1 | 3 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 3 | 5
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 17 | 14 | 16 [14 to 17] | 16 [14 to 17]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4
  Male | 0 | 0 | 1 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Convergence Insufficiency Symptom Survey
Description: This survey quantifies convergence insufficiency symptoms on a scale. The scale measures the severity of symptoms from the condition, convergence insufficiency. Score on a scale can range from 0 (least) to 60 (worst). This survey has been proven to be an effective and accurate gauge by previous research and study groups.
Time Frame: Assessed up to 12 months
Population: All participants met the criteria of the study
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Single Vision Glasses | Single Vision Glasses With Anti-glare Coating | Eyezen
Number analyzed (Participants) | 1 | 1 | 1
score on a scale | 29 (0) | 22 (0) | 14 (0)

2. Secondary Outcome: Convergence Breaking Point at Near (Base Out Prism)
Description: This outcome measurement was the maximum base out prism diopters when the patient first reported diplopia of a near target or started suppressing one of the eyes as determined by the examiner.
Time Frame: Assessed up to 12 months
Population: All participants meet inclusion criteria. However, 2 of the 5 participants did not return for the follow up visit and therefore do not have outcome measurements.
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Single Vision Glasses | Single Vision Glasses With Anti-glare Coating | Eyezen
Number analyzed (Participants) | 1 | 1 | 1
prism diopters | 16 (0) | 40 (0) | 12 (0)

ADVERSE EVENTS:
Time Frame: Each participant was enrolled for roughly 3 months and was able to keep the glasses after that period.
Description: The definitions did not differ.
Arm/Group | Single Vision Glasses | Single Vision Glasses With Anti-glare Coating | Eyezen
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-04-02): https://cdn.clinicaltrials.gov/large-docs/22/NCT03123822/Prot_003.pdf